CLINICAL TRIAL: NCT01500226
Title: Phase 3, Multicenter, Randomized, Double Blind, Active-Controlled Study of the Safety and Efficacy of Rolapitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) in Subjects Receiving Moderately Emetogenic Chemotherapy
Brief Title: Ph 3 Safety/Efficacy Study of Rolapitant for Prevention of CINV in Subjects Receiving Moderately Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TS-P04834
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2014-07

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Rolapitant; Nausea; Vomiting; CINV; Chemotherapy
MeSH Terms: conditions — Vomiting; Nausea | interventions — rolapitant; Granisetron; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo + Granisetron + Dexamethasone (Placebo Comparator): Day 1: Placebo + Granisetron (2 mg PO)+ Dexamethasone (20 mg PO) Days 2-3: Granisetron (2 mg PO) will be administered orally.
  Interventions: Drug: Granisetron; Drug: Dexamethasone; Drug: Placebo
- Rolapitant (Experimental): Day 1: Rolapitant (200 mg PO) + Granisetron (2 mg PO)+ Dexamethasone (20 mg PO) Days 2-3: Granisetron (2 mg PO) will be administered orally.
  Interventions: Drug: Rolapitant; Drug: Granisetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Rolapitant — (4 X 50 mg capsule) 200 mg PO
  Other Names: Varubi
  Arms: Rolapitant
Drug: Granisetron — 2 mg PO
  Other Names: Kytril; Granisol
Drug: Dexamethasone — 20 mg PO
  Other Names: Decadron
Drug: Placebo — (4 X 0 mg capsules) 0 mg PO
  Other Names: Placebo to match Rolapitant
  Arms: Placebo + Granisetron + Dexamethasone

SUMMARY:
This is a Phase 3, multicenter, randomized, parallel-group, double-blind, active-controlled study of rolapitant in subjects receiving MEC. Rolapitant or placebo will be administered prior to the initiation of chemotherapy on Day 1 with granisetron and dexamethasone. Subjects will record all events of emesis and the use of rescue medication for established nausea and/or vomiting, and will indicate the severity of nausea they experienced in each of the previous 24 hours in the Nausea and Vomiting (NV) Subject Diary prior to the MEC administration through Day 6 in Cycle 1. Health-related quality of life will be measured by the FLIE Questionnaire on Day 6 of Cycle 1. Safety and tolerability will be assessed by clinical review of adverse events (AEs), physical examination, electrocardiograms (ECGs), and safety laboratory values. All subjects are expected to complete Cycle 1 and will have the option of participating in up to five additional cycles.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, parallel-group, double-blind, active-controlled study of rolapitant in subjects receiving MEC. Rolapitant or placebo will be administered orally 1-2 hours prior to the initiation of chemotherapy on Day 1. Granisetron (2 mg PO) and dexamethasone (20 mg PO) will be administered approximately 30 minutes before initiation of chemotherapy. Subjects will continue to receive granisetron (2 mg daily) on Days 2 and 3. Subjects will record all events of emesis and the use of rescue medication for established nausea and/or vomiting, and will indicate the severity of nausea they experienced in each of the previous 24 hours in the Nausea and Vomiting (NV) Subject Diary prior to the MEC administration through Day 6 in Cycle 1. Health-related quality of life will be measured by the FLIE Questionnaire on Day 6 of Cycle 1. Safety and tolerability will be assessed by clinical review of adverse events (AEs), physical and neurological examinations, vital signs, electrocardiograms (ECGs), and safety laboratory values including BUN and creatinine. All subjects are expected to complete Cycle 1 and will have the option of participating in up to five additional cycles. Blood samples may be collected and stored in this study and may be analyzed for future biomarker research related to safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, of either gender, and of any race
* Naïve to moderately or highly emetogenic chemotherapy, and is to receive a first course of MEC including one or more of the following agents: cyclophosphamide IV (<1500 mg/m2), doxorubicin, epirubicin, carboplatin, idarubicin, ifosfamide, irinotecan, daunorubicin, cytarabine IV (>1 g/m2).
* Karnofsky performance score of ≥60
* Predicted life expectancy of ≥4 months
* Adequate bone marrow, kidney, and liver function

Exclusion Criteria:

* Contraindication to the administration of prescribed MEC agent,granisetron, or dexamethasone
* Is pregnant or breast feeding
* Has taken the following agents within the last 48 hours 5-HT3 antagonists,Phenothiazines,Benzamides,Domperidone,Cannabinoids,NK1 antagonist, Benzodiazepines
* Scheduled to receive any other chemotherapeutic agent with an emetogenicity level of 3 or above (Hesketh Scale) from Day -2 through Day 6, except on Day 1
* Scheduled to receive any radiation therapy to the abdomen or pelvis from Day -5 through Day 6
* Has received systemic corticosteroids or sedative antihistamines within 72 hours of Day 1 of the study except as premedication for chemotherapy (e.g., taxanes)
* Symptomatic primary or metastatic CNS disease.
* Has ongoing vomiting, retching, clinically significant nausea caused by any etiology, or has a history of anticipatory nausea and vomiting.
* Has vomited and/or has had dry heaves/retching within 24 hours prior to the start of MECon Day 1 in Cycle 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1369 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vargo, MD, Study Director — Tesaro, Inc.
Locations (1):
- TESARO Inc, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Schwartzberg LS, Modiano MR, Rapoport BL, Chasen MR, Gridelli C, Urban L, Poma A, Arora S, Navari RM, Schnadig ID. Safety and efficacy of rolapitant for prevention of chemotherapy-induced nausea and vomiting after administration of moderately emetogenic chemotherapy or anthracycline and cyclophosphamide regimens in patients with cancer: a randomised, active-controlled, double-blind, phase 3 trial. Lancet Oncol. 2015 Sep;16(9):1071-1078. doi: 10.1016/S1470-2045(15)00034-0. Epub 2015 Aug 10. PMID 26272768

RESULTS

PARTICIPANT FLOW:
Groups:
- Rolapitant + Granisetron + Dexamethasone: * Oral dose of rolapitant 180 mg (equivalent to 200mg rolapitant hydrochloride monohydrate) 1-2 h before administration of chemotherapy.
  * Granisetron (2 mg orally) about 30 min before chemotherapy. Subsequently, granisetron 2mg was administered orally to all patients once daily on days 2-3
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy.
- Placebo + Granisetron + Dexamethasone: * Matching placebo 1-2 h before administration of chemotherapy
  * Granisetron (2 mg orally) about 30 min before chemotherapy. Subsequently, granisetron 2mg was administered orally to all patients once daily on days 2-3
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy
Period: Overall Study
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Started | 684 (Number of randomized patients) | 685
Completed | 185 (Number of patients who completed 6 cycles) | 191
Not Completed | 499 | 494
Not completed — Adverse Event | 31 | 38
Not completed — Chemo Completed or Change in Therapy | 235 | 237
Not completed — Withdrawal by Subject | 93 | 96
Not completed — Death | 12 | 4
Not completed — Disease Progression | 16 | 14
Not completed — Protocol Violation | 53 | 39
Not completed — Physician Decision | 17 | 15
Not completed — Lack of Efficacy | 14 | 30
Not completed — Lost to Follow-up | 9 | 5
Not completed — Other Reasons | 19 | 16

BASELINE CHARACTERISTICS:
Population: * 684 subjects were randomized to Rolapitant and 685 were randomized to control;
  * 670 of those randomized to Rolapitant received study drug in C1; 674 of those who were randomized to control received study drug in C1.
  * 4 Rolapitant subject and 8 control subject were from GCP-non-compliant sites.
  * MITT = 666 Rolapitant and 666 control
Groups:
- Rolapitant + Granisetron + Dexamethasone: * Oral dose of rolapitant 180 mg (equivalent to 200 mg rolapitant hydrochloride monohydrate) 1-2 h before administration of chemotherapy
  * Granisetron (2 mg orally) about 30 min before chemotherapy. Subsequently, granisetron 2mg was administered orally to all patients once daily on days 2-3
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy
- Total: Total of all reporting groups
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone | Total
Number analyzed (Participants) | 666 | 666 | 1332
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (11.65) | 56.6 (12.01) | 56.7 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 531 | 536 | 1067
  Male | 135 | 130 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77 | 70 | 147
  Not Hispanic or Latino | 584 | 593 | 1177
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 92 | 84 | 176
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 24 | 29 | 53
  White | 508 | 512 | 1020
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: No Emetic Episodes and No Rescue Medication
Description: The primary objective of this study is to determine whether administration of rolapitant with granisetron and dexamethasone improves CINV in the delayed phase (>24 to 120 hours) of CINV compared with administration of placebo with granisetron and dexamethasone in subjects receiving MEC. The primary outcome will be based on complete response (defined as no emesis and no rescue medication) in the delayed phase (>24 to 120 hours).
Time Frame: >24 to 120 hours post chemotherapy
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Number analyzed (Participants) | 666 | 666
percentage of particpants | 71.3 [67.7 to 74.7] | 61.6 [57.7 to 65.3]
Statistical Analysis 1: Comparison: Rolapitant + Granisetron + Dexamethasone vs Placebo + Granisetron + Dexamethasone; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — To control for multiplicity, analyses were performed hierarchically. For the CR delayed the threshold for statistical significance was 0.05; no further adjustment for multiplicity were required for the primary endpoint; Cochran Mantel Haenszel (CMH) test was stratified by sex. Missing data were imputed as treatment failures; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.2 to 2.0]

2. Secondary Outcome: Acute Phase Response
Description: To determine the effect of rolapitant on complete response rates in the acute (0 to 24 hours) phase of CINV.
Time Frame: 0 to 24 hours
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Number analyzed (Participants) | 666 | 666
percentage of participants | 83.5 [80.4 to 86.2] | 80.3 [77.1 to 83.3]
Statistical Analysis 1: Comparison: Rolapitant + Granisetron + Dexamethasone vs Placebo + Granisetron + Dexamethasone; Test type: Superiority or Other; p = 0.143, Cochran-Mantel-Haenszel — To control for multiplicity, analyses were performed hierarchically. CR-acute was tested only if the result for the primary endpoint, CR delayed, was statistically significant; Cochran Mantel Haenszel (CMH) test was stratified by sex. Missing data were imputed as treatment failures; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.9 to 1.6]

3. Secondary Outcome: Overall Response Rate
Description: To determine the effect of rolapitant on complete response rate in the overall (0 to 120 hours) phase of CINV.
Time Frame: 0 to 120 hours
Population: MITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Number analyzed (Participants) | 666 | 666
percentage of participants | 68.6 [64.9 to 72.1] | 57.8 [54.0 to 61.6]
Statistical Analysis 1: Comparison: Rolapitant + Granisetron + Dexamethasone vs Placebo + Granisetron + Dexamethasone; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — To control for multiplicity, analyses were performed hierarchically. CR overall was tested only if both CR delayed and CR acute were statistically significant; Cochran Mantel Haenszel (CMH) test was stratified by sex. Missing data were imputed as treatment failures; Odds Ratio (OR) = 1.6, 95% CI 2-sided [1.3 to 2.0]

ADVERSE EVENTS:
Time Frame: Up to 6 cycles (median number of cycles=4; median duration of each cycle = 21 days) of treatment
Groups:
- Rolapitant + Granisetron + Dexamethasone: * Oral dose of rolapitant 180 mg (equivalent to 200 mg rolapitant hydrochloride monohydrate) 1-2 h before administration of chemotherapy
  * Granisetron (2 mg orally) about 30 min before chemotherapy. Subsequently, granisetron 2mg was administered orally to all patients once daily on days 2-3
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy
    * 684 subjects were randomized to Rolapitant
    * 670 of those randomized to Rolapitant received rolapitant in C1
    * Safety = 670 Rolapitant
- Placebo + Granisetron + Dexamethasone: * Matching placebo 1-2 h before administration of chemotherapy
  * Granisetron (2 mg orally) about 30 min before chemotherapy. Subsequently, granisetron 2mg was administered orally to all patients once daily on days 2-3
  * Dexamethasone (20 mg orally) about 30 min before chemotherapy
    * 685 subjects were randomized to control
    * 674 of those who were randomized to control received control in C1
    * Safety = 674 control
Arm/Group | Rolapitant + Granisetron + Dexamethasone | Placebo + Granisetron + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 89/670 | 103/674
Other Adverse Events (participants affected / at risk) | 540/670 | 542/674
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rolapitant + Granisetron + Dexamethasone (N=670) | Placebo + Granisetron + Dexamethasone (N=674)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 14 | 25
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 7 | 13
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 2 | 4
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 1
Jejunal Perforation (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Disease Progression (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Catheter Site Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Device Related Sepsis (Infections and infestations) | 1 | 0
Diarrhoea Infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 1
Fungaemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 4 | 2
Oral Fungal Infection (Infections and infestations) | 1 | 0
Pelvic Infection (Infections and infestations) | 0 | 1
Peridiverticular Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Postoperative Wound Infection (Infections and infestations) | 1 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
C-Reactive Protein Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 3 | 4
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cerebral Haematoma (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 1 | 0
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Skin Erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 0
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 3
Thrombosis (Vascular disorders) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rolapitant + Granisetron + Dexamethasone (N=670) | Placebo + Granisetron + Dexamethasone (N=674)
Anaemia (Blood and lymphatic system disorders) | 67 | 50
Leukopenia (Blood and lymphatic system disorders) | 37 | 31
Neutropenia (Blood and lymphatic system disorders) | 96 | 84
Abdominal Pain (Gastrointestinal disorders) | 34 | 31
Constipation (Gastrointestinal disorders) | 114 | 138
Diarrhoea (Gastrointestinal disorders) | 92 | 101
Dyspepsia (Gastrointestinal disorders) | 46 | 42
Nausea (Gastrointestinal disorders) | 76 | 97
Stomatitis (Gastrointestinal disorders) | 40 | 46
Vomiting (Gastrointestinal disorders) | 14 | 39
Asthenia (General disorders) | 78 | 78
Fatigue (General disorders) | 179 | 183
Mucosal Inflammation (General disorders) | 41 | 30
Urinary Tract Infection (Infections and infestations) | 57 | 45
Decreased Appetite (Metabolism and nutrition disorders) | 92 | 87
Dehydration (Metabolism and nutrition disorders) | 25 | 37
Hypomagnesaemia (Metabolism and nutrition disorders) | 41 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 34
Bone Pain (Musculoskeletal and connective tissue disorders) | 42 | 40
Dizziness (Nervous system disorders) | 69 | 71
Dysgeusia (Nervous system disorders) | 29 | 38
Headache (Nervous system disorders) | 82 | 109
Insomnia (Psychiatric disorders) | 32 | 55
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 37
Alopecia (Skin and subcutaneous tissue disorders) | 157 | 172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No